CLINICAL TRIAL: NCT06673927
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics of YZJ-1139 in Healthy Participants
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Doses of YZJ-1139 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Haiyan Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YZJ-1139-1-01
Record Dates: First submitted 2024-11-01; First posted 2024-11-05 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-11

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Dose escalation
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YZJ-1139 Single-dose Group (Experimental): Subjects will be randomized into two groups： the experimental group will receive YZJ-1139; the control group will receive placebo.
  Interventions: Drug: YZJ-1139
- YZJ-1139 multiple-dose Group (Experimental): Subjects will be randomized into two groups；the experimental group will receive YZJ-1139; the control group will receive placebo once a day, 7 days.
  Interventions: Drug: YZJ-1139; Drug: Placebo

INTERVENTIONS:
Drug: YZJ-1139 — Single oral dose, 2mg, 5mg, 10mg, 20mg, 40mg, 60mg, 80mg
  Arms: YZJ-1139 Single-dose Group
Drug: YZJ-1139 — Multiple Dosing ，Each oral dose of 10 mg，20 mg，40 mg or 60 mg
  Arms: YZJ-1139 multiple-dose Group
Drug: Placebo — Placebo administration
  Arms: YZJ-1139 multiple-dose Group

SUMMARY:
Primary Objective：

1. To evaluate the tolerability, safety of single and multiple doses of YZJ-1139 in healthy participants
2. To evaluate the pharmacokinetic of single and multiple doses of YZJ-1139 in healthy participants

Secondary objectives:

To explore the safe tolerated dose of YZJ-1139, provide data support for the design of phase II dosing regimen

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects, with the proportion of a single gender in each group not less than 1/3;
2. Aged between 18 and 45 years (inclusive of 18 and 45 years);
3. The body mass index (BMI) ranges from 19 to 24 (inclusive of 19 and 24), where BMI = weight (kg) / height squared (m²). At the time of entering the study, the weight of female volunteers must be no less than 50 kg, and that of male volunteers must be no less than 55 kg;
4. Those who pass comprehensive physical examinations (vital signs, height, weight, and chest and abdominal examinations, etc.) and laboratory tests (blood routine, blood biochemistry, urine routine, electrocardiogram, infectious disease screening, etc.), and have no abnormalities or only minor abnormalities without clinical significance in 12-lead electrocardiogram, abdominal B-ultrasound (liver, gallbladder, pancreas, spleen, and kidneys), anteroposterior and lateral chest radiographs, etc.;
5. Volunteers who can comprehend the procedures and methods of this study, are willing to strictly adhere to the clinical trial protocol to complete the trial, and sign the informed consent form.

Exclusion Criteria:

1. After researchers determine that the subject has a disease that affects drug absorption, distribution, metabolism, and excretion or may reduce compliance (cardiovascular, liver, kidney, gastrointestinal, immune, hematological, endocrine, metabolic, cancer, psychiatric and neurological conditions);
2. A history of specific allergic reactions (such as asthma, eczema, allergic dermatitis); known allergies to the trial drug and its excipient components; a history of drug allergies;
3. A history of obstructive sleep apnea or chronic obstructive pulmonary disease;
4. A history of severe unconscious hypoglycemia;
5. A history of stroke, chronic epilepsy, or neurological disorders;
6. A history of diminished memory or abnormal behavior;
7. A history of drug dependence within the past 2 years (smoking excluded), seizure disorders, syncope history;
8. A clinically significant illness within the past month before enrollment, especially severe infections, trauma, or major surgery;
9. The use of any prescription drugs or herbal medicines within the past month before enrollment, and non-prescription drugs or food supplements within the past 2 weeks;
10. Regular use of sedatives, sleeping pills, or other addictive drugs, and positive urine drug screening;
11. had donated blood within the 3 months prior to the study, or had severe blood loss equivalent to at least 500 mL of blood loss;
12. Hepatitis B surface antigen positive, hepatitis C antibody positive, HIV antibody positive, syphilis antibody positive;
13. Patients who took CYP3A enzyme inhibitors (itraconazole, erythromycin, boprevir, etc.), CYP3A enzyme inducers (rifampicin, carbamazepine) and/or CNS inhibitors (benzodiazepines, opioids, tricyclic antidepressants, etc.) 2 weeks before inclusion;
14. Have a history of alcohol abuse (drinking 14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or about 100 ml of wine) and test positive for alcohol;
15. Smokers who smoked more than 5 or equivalent cigarettes per day in the 3 months before the test and those who tested positive for nicotine should not give up smoking during the test;
16. Drinking excessive tea and coffee drinks (more than 8 cups) per day;
17. Drinking alcohol, eating food and drink rich in xanthine or caffeine (including chocolate, tea, coffee, cola, etc.) or eating grapefruit, limes, etc., or food and drink prepared from them in the 3 days prior to inclusion;
18. Participated in any clinical drug research or clinical trial of medical device within 3 months prior to screening;
19. Pregnant and lactating women within 6 months from the subject's signature to the last administration of the study drug; Fertile women who do not use effective non-hormonal contraception (Iuds, barrier contraception with spermicide or surgical sterilization, etc.) or are unwilling to continue using these methods; Fertile men are reluctant to use physical methods of contraception; Women who were menstruating during the trial (see annex 3 for details);
20. There are any subjects that the investigator considers unsuitable for participation in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 to Day 3 post single dose；From Day 1 to Day 14 post multiple dose；

SECONDARY OUTCOMES:
Cmax of YZJ-1139 | From Day 1 to Day 2 post single dose；From Day 1 to Day 8 post multiple dose
  Cmax is defined as the maximum concentration of drug.
AUCinf of YZJ-1139 | From Day 1 to Day 2 post single dose；From Day 1 to Day 8 post multiple dose
  AUCinf is defined as the concentration of drug extrapolated to infinite time.
AUClast of YZJ-1139 | From Day 1 to Day 2 post single dose；From Day 1 to Day 8 post multiple dose
  AUClast is defined as the concentration of drug from time zero to the last observable concentration.
AUC0-τ of YZJ-1139 | From Day 1 to Day 8 post multiple dose
  AUC0-τ is defined as the area under the concentration-time curve over the dosing interval
Css,avg of YZJ-1139 | From Day 1 to Day 8 post multiple dose
  Css,avg is defined as the average steady state concentration
Css,min of YZJ-1139 | From Day 1 to Day 8 post multiple dose
  Css,min is defined as the minimum observed concentration at steady
Tmax of YZJ-1139 | From Day 1 to Day 2 post single dose；From Day 1 to Day 8 post multiple dose
  Tmax is defined as the time (observed time point) of Cmax
t1/2 of YZJ-1139 | From Day 1 to Day 2 post single dose；From Day 1 to Day 8 post multiple dose
CL/F of YZJ-1139 | From Day 1 to Day 2 post single dose；From Day 1 to Day 8 post multiple dose
  CL/F is defined as the apparent oral clearance following administration of the drug
Vz/F of YZJ-1139 | From Day 1 to Day 2 post single dose；From Day 1 to Day 8 post multiple dose
  Vz/F is defined as the apparent volume of distribution of the drug
Rac of YZJ-1139 | From Day 1 to Day 8 post multiple dose
  Rac is defined as the accumulation Ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Ditan Hospital Capital Medical University, Beijing, China